CLINICAL TRIAL: NCT05980169
Title: The Effect of Low Frequency Soundwave Stimulation on Chemotherapy Induced Peripheral Neuropathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCC-23-021
Record Dates: First submitted 2023-07-10; First posted 2023-08-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-01

CONDITIONS: Gynecologic Cancer; Neuropathy;Peripheral
Keywords: Chemotherapy; Neuropathy; Soundwave Stimulation
MeSH Terms: conditions — Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort A (Experimental): In this arm, patients with newly diagnosed gynecologic cancer starting chemotherapy treatment with carboplatin and paclitaxel will receive up to 8 cycles of SensoniQ treatment along with their chemotherapy (weekly or every 21 days depending on the regimen).
  Interventions: Device: SensoniQ Treatment Station
- Cohort B (Experimental): Cohort B was closed on April 1st, 2025 due to not meeting the 30% improvement CIPNS objective. Enrollment was closed for Cohort B and all maintenance treatment and follow-ups were discontinued. No safety issues were identified during data analysis. In this arm, gynecologic cancer patients with persistent neuropathy following treatment with platinum agent and paclitaxel will receive a 30-minute SensoniQ treatment twice weekly for 4 weeks.
  Interventions: Device: SensoniQ Treatment Station

INTERVENTIONS:
Device: SensoniQ Treatment Station — The SensoniQ® Treatment Station is a chemotherapy chair with multiple transducers that release low- frequency sound waves to different points on the body in a preset frequency, distribution and time during a chemotherapy infusion.
  Other Names: Wave Chair

SUMMARY:
The goal of this clinical trial is to assess the efficacy of SensoniQ® Treatment Station in preventing or reducing chemotherapy induced peripheral neuropathy symptoms (CIPNS) in patients receiving frontline carboplatin and paclitaxel chemotherapy for a gynecologic malignancy. This study will also assess the improvement of CIPNS in patients who have previously received carboplatin and paclitaxel therapy with persistent Grade 2 or worse neuropathy.

The main questions this clinical trial aims to answer are:

1. To investigate the efficacy of SensoniQ® Treatment Station on the prevention or reduction of CIPNS in gynecologic oncology patients receiving front line carboplatin and paclitaxel.
2. To investigate the efficacy of SensoniQ® Treatment Station on the improvement of existing CIPNS in patients who previously received chemotherapy with platinum agent and paclitaxel for a gynecologic malignancy

DETAILED DESCRIPTION:
Chemotherapy induced neuropathy symptoms (CIPNS) are a common side effect in patients undergoing treatment for gynecologic malignancies. The most common treatment is a combination of paclitaxel and carboplatin. A previous analysis of these patients show that 71% experience chemo induced peripheral with neuropathy with 30% experiencing Grade 2 and 32% experiencing Grade 3. There is currently no intervention to prevent CIPNS and only one medication, duloxetine, is recommended as treatment based on ASCO guidelines.

The SensoniQ® Treatment Station is a chemotherapy chair with multiple transducers that release low- frequency sound waves to different points on the body in a preset frequency, distribution and time during a chemotherapy infusion. Previous investigational studies using SensoniQ® Treatment during chemotherapy infusion showed a reduction in neuropathy without any additional side effects or complications.

This study seeks to show patient response measured by questionnaires to SensoniQ® Treatment and correlate with neurologic test findings to show reduced CIPNS in patients undergoing frontline chemotherapy with carboplatin and paclitaxel as well as improvement in patients with existing CIPNS. This treatment has the potential to change recommendations for prevention of CIPNS and improve adherence to treatment and quality of life.

ELIGIBILITY:
Inclusion Criteria: Patients must meet all the following inclusion criteria to be eligible for inclusion in the study:

1. Patients must be age 18 or older.
2. Histologically confirmed gynecologic malignancy.
3. Eastern Cooperative Oncology Group performance status of 0 to 2.
4. Be willing and able to participate in all required evaluations for the protocol
5. Speak, read, and understand English

   Cohort A patients must have:
6. Carboplatin and paclitaxel prescribed as first line treatment. Patients may also receive Trastuzumab, Bevacizumab, Pembrolizumab or Dostarlimab in conjunction with carboplatin and paclitaxel as these regimens are standard of care for specific cancers. Additional drugs may be acceptable after review and approval by the PI. In the event of a hypersensitivity reaction with paclitaxel, subjects may be switched to docetaxel and continue on study. In the event of a carboplatin hypersensitivity reaction, additional drugs or alterations to the treatment regimen may be changed after review and approval by the PI.

Cohort B patients must have:

7. Received prior treatment with a platinum agent and paclitaxel with a persistent CTCAE defined Grade 2 or worse neuropathy

-

Exclusion Criteria: Patients with any of the following will not be included in the study:

1. Current diagnosis of comorbidity causing neuropathy (including peripheral vascular disease, lupus, Sjogren's syndrome, rheumatoid arthritis). Patients with diabetes may participate if baseline exam is negative for neuropathy symptoms and HbA1c < 7.
2. Pregnant
3. DVT diagnosed within 4 weeks prior to treatment
4. Body weight greater 195kg

Cohort A patients:

6. Previous treatment with taxane therapy 7. Preexisting diagnosis of neuropathy 8. Currently prescribed gabapentin, duloxetine or pregabalin

Cohort B patients:

9. Diagnosis of neuropathy prior to cancer treatment

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study protocol is specific to gynecological oncology studies. The study only applies to female patients.
Enrollment: 80 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
FACT/GOG-NTX & EORTC QLQ-CIPN20 | 18 months
  Percent of patients reporting neuropathy based on post treatment Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity Questionnaire (FACT/GOG NTX) and European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-CIPN Twenty Item Subscale (EORTC QLQ-CIPN20) scores (This primary outcome is specific to Cohort A)
FACT/GOG-NTX & EORTC QLQ CIPN-20 | 18 months
  Percent reduction in neuropathy based on post treatment FACT/GOG NTX and EORTC QLQ-CIPN 20 score compared to pretreatment score (This primary outcome measure is specific to Cohort B).

SECONDARY OUTCOMES:
Neurologic Exams | 18 months
  Change in score from pretreatment to post-treatment neurologic exams (Specific to both cohorts A & B).
FACT/GOG NTX & EORTC QLQ-CIPN 20 | 18 months
  Direct correlation of FACT/GOG NTX and EORTC QLQ-CIPN 20 scores to non-invasive neurologic scores (Specific to both cohorts A & B).
Safety & Tolerability | 18 months
  Safety and tolerability based on AEs & SAEs related to the device (to both cohorts A & B).
Dose of chemotherapy | 18 months
  Total dose of chemotherapy (Specific to cohort A).
Overall Response Rate | 18 months
  ORR at 6 months post treatment per FACT/GOG NTX and EORTC QLQ-CIPN 20 scores and non-invasive neurologic test scores (specific to cohort B).
FACT/GOG NTX & EORTC QLQ-CIPN20 maximum reduction | 18 months
  Assess FACT/GOG NTX and EORTC QLQ-CIPN20 scores at specified visits to determine the treatment number at which maximum reduction from baseline score is reported (specific to cohort B).
Treatment Completion | 18 months
  Time for treatment completion (Specific to cohort A).
Sustained Response Assessment | 18months
  • Assess sustained response to treatment in patients who received 8 treatments versus patients who received 8 treatments with 6 maintenance treatments

CONTACTS AND LOCATIONS:
Locations (1):
- James T Sonnenberg, Augusta, Georgia, United States